CLINICAL TRIAL: NCT05817760
Title: Evaluation of Z-plasty Versus Heineke-Mikulicz Scrotoplasty in the Management of Penoscrotal Web in Pediatric Age Group
Brief Title: Z-plasty and Heineke-Mikulicz Scrotoplasty in the Management of Penoscrotal Web
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egyptian Biomedical Research Network (Network)
Responsible Party: Principal Investigator, Ahmed Elrouby, Associate Professor of pediatric Surgery, Egyptian Biomedical Research Network
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0305354
Record Dates: First submitted 2023-03-19; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Urologic Diseases
Keywords: Penoscrotal web; Z-scrotoplasty; Heineke-Mikulicz
MeSH Terms: conditions — Urologic Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Z-scrotoplasty (Experimental): Pediatric patients with congenital penoscrotal web who will be treated by Z-scrotoplasty
  Interventions: Procedure: Z-scrotoplasty
- Heineke-Mikulicz scrotoplasty (Experimental): Pediatric patients with congenital penoscrotal web who will be treated by Heineke-Mikulicz scrotoplasty
  Interventions: Procedure: Heineke-Mikulicz scrotoplasty

INTERVENTIONS:
Procedure: Z-scrotoplasty — Z shape incision of the penoscrotal web and closure
  Arms: Z-scrotoplasty
Procedure: Heineke-Mikulicz scrotoplasty — Transverse incision of the penoscrotal web with vertical closure
  Arms: Heineke-Mikulicz scrotoplasty

SUMMARY:
The goal of this clinical trial is to compare the surgical outcome of Z-scrotoplasty versus Heineke-Mikulicz scrotoplasty in the management of congenital penoscrotal web in pediatric age group.

The main question[s] it aims to answer are:

• Question 1: Is there a difference in the surgical outcome between using Z-scrotoplasty and Heinke Miculickz scrotoplasty in the management of congenital penoscrotal web?] Participants will be divided into two groups; Group A treated by Z-scrotoplasty and Group B treated by Heineke Miculickz scrotoplasty.

DETAILED DESCRIPTION:
Background: The penoscrotal web may be congenital or acquired after excessive removal of ventral skin during circumcision. There are several previously described surgical techniques for the treatment of congenital webbed penis without a clear comparison between their outcomes. Purpose: the objective of our study was to compare the surgical results of Z-scrotoplasty and Heineke-Mikulicz scrotoplasty in the treatment of congenital webbed penis. Patients & Methods: Our prospective study included 40 uncircumcised patients presented with a webbed penis. They were divided into group A which was treated by Z-scrotoplasty and group B which was treated by Heineke-Mikulicz scrotoplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients with congenital penoscrotal web in the pediatric age group

Exclusion Criteria:

* Patients with any penile anomalies

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Number of patients who developed post-operative penile edema, hematoma, adequate skin coverage and wound contracture with recurrent webbing will be assessed | One post-operative year
  Post-operative follow up for the detection of penile edema, hematoma, skin coverage and the development of any wound contracture and consequently recurrent webbing

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elrouby, MD, Study Director — Pediatric Surgery department
Locations (1):
- Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elrouby A. Evaluation of Z-plasty versus Heineke-Mikulicz scrotoplasty in the management of penoscrotal web in pediatric age group. BMC Urol. 2024 Mar 22;24(1):66. doi: 10.1186/s12894-024-01450-7. PMID 38519937